CLINICAL TRIAL: NCT02620020
Title: A Randomized, Double-blind, Multi-dose, Placebo-controlled Phase 2/3 Study to Evaluate the Efficacy and Safety of Fasinumab in Patients With Moderate to Severe Chronic Low Back Pain
Brief Title: A Study to Determine the Efficacy and Safety of Fasinumab for the Treatment of Adults With Chronic Low Back Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R475-PN-1524; 2015-003782-28 (EudraCT Number)
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — fasinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fasinumab 6 mg SC Q4W and Placebo IV Q8W (Experimental): Participants randomized to the fasinumab 6 mg SC Q4W arm received fasinumab 12 mg SC on Day 1 (loading dose) and then 6 mg SC (planned maintenance dose) at Weeks 4, 8, and 12 for a total of 4 doses. Matching placebo was received via intravenous (IV) infusion Q8W on Day 1 and at Week 8.
  Interventions: Drug: Fasinumab; Drug: placebo
- Fasinumab 9 mg SC Q4W and Placebo IV Q8W (Experimental): Participants randomized to the fasinumab 9 mg SC Q4W arm received 18 mg SC on day 1 (loading dose) and then 9 mg SC (planned maintenance dose) at weeks 4, 8, and 12 for a total of 4 doses. Matching placebo IV Q8W was received on Day 1 and at Week 8.
  Interventions: Drug: Fasinumab; Drug: placebo
- Fasinumab 9 mg IV Q8W and Placebo SC Q4W (Experimental): Participants randomized to the fasinumab 9 mg IV Q8W arm received IV infusions of fasinumab 9 mg on Day 1 and Week 8, for a total of 2 doses. Matching placebo SC Q4W was received on day 1 and at weeks 4, 8, and 12.
  Interventions: Drug: Fasinumab; Drug: placebo
- Placebo SC Q4W and Placebo IV Q8W (Experimental): Participants randomized to the matching placebo subcutaneously (SC) every four weeks (Q4W) arm received SC placebo in a manner similar to the SC loading dose of the active groups (placebo loading dose) on Day 1 and then an SC injection of placebo at weeks 4, 8, and 12 for a total of 4 doses. Matching placebo intravenously (IV) every 8 weeks (Q8W) was received on Day 1 and at Week 8.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Fasinumab — Participants received fasinumab SC or IV, Q4W or Q8W.
  Other Names: REGN475
  Arms: Fasinumab 6 mg SC Q4W and Placebo IV Q8W; Fasinumab 9 mg IV Q8W and Placebo SC Q4W; Fasinumab 9 mg SC Q4W and Placebo IV Q8W
Drug: placebo — Participants received placebo matching to fasinumab SC or IV, Q4W or Q8W.

SUMMARY:
The main objective of the trial is to evaluate the efficacy of fasinumab compared to placebo as measured by the change from baseline in the average daily Low Back Pain Intensity (LBPI) Numerical Rating Scale (NRS).

Secondary objectives of the study are to evaluate the efficacy of fasinumab compared to placebo as measured by:

* Change from baseline in the Roland Morris disability questionnaire (RMDQ) total score
* Change from baseline in the Patient Global Assessment (PGA) of Low Back Pain (LBP) score
* Change from baseline in the average daily LBPI NRS score

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female ≥35 years of age at the screening visit
2. Clinical diagnosis of chronic moderate to severe LBP (nonradiculopathic)for ≥3 months
3. History of regular analgesic medication
4. History of inadequate pain relief or intolerance to analgesics used for chronic LBP
5. Willing to discontinue current pain medication

Key Exclusion Criteria:

1. History of lumbosacral radiculopathy within the past 2 years
2. Evidence on baseline lumbar spine magnetic resonance imaging of potentially confounding conditions
3. Recent use of longer acting pain medications
4. Evidence of destructive arthropathy
5. Other medical conditions that may interfere with participation or accurate assessments during the trial

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2017-02-03 (Actual); Study Completion 2017-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (74):
- United States (58):
  - Birmingham, Alabama
  - Chandler, Arizona
  - Glendale, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Carlsbad, California
  - Lakewood, California
  - Long Beach, California
  - Sacramento, California
  - San Diego, California
  - Santa Rosa, California
  - Vista, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Littleton, Colorado
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Fort Myers, Florida
  - Leesburg, Florida
  - Miami, Florida
  - Orlando, Florida
  - Chicago, Illinois
  - Evansville, Indiana
  - Council Bluffs, Iowa
  - Worcester, Massachusetts
  - Edina, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Elkhorn, Nebraska
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Jamaica, New York
  - New York, New York
  - Williamsville, New York
  - Cary, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Duncansville, Pennsylvania
  - Anderson, South Carolina
  - Greer, South Carolina
  - Bristol, Tennessee
  - Knoxville, Tennessee
  - Cypress, Texas
  - Dallas, Texas
  - Lubbock, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
- Canada (2):
  - London, Ontario
  - Toronto, Ontario
- Czechia (2):
  - Prague
  - Rychnov nad Kněžnou
- Denmark (2):
  - Aalborg
  - Ballerup Municipality
- Tallinn, Estonia
- Hungary (3):
  - Budapest
  - Gyula
  - Szolnok
- Poland (6):
  - Bialystok
  - Lodz
  - Lublin
  - Rzeszów
  - Warsaw
  - Zgierz

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 105 sites in US, CA & EU from 26Jan2016 - 13Sep2017. Of 1,783 participants screened, 563 randomized to 1 of 4 groups stratified by baseline low back pain numerical rating scale (LBP NRS) score (<7, ≥7), duration of chronic LBP (<5, ≥5yrs) & max. Kellgren-Lawrence (K-L) score (≤2, >2) at any knee/ hip joint at screening.
Pre-assignment Details: The study consisted of a screening period of up to 30 days & a 7-day pre-randomization period during which pain medication, except study-provided rescue medication, was discontinued. Confirmation of no exclusionary findings on joint on which imaging was performed during screening must have been received before a participant could be randomized.
Period: Overall Study
Arm/Group | Placebo SC Q4W and Placebo IV Q8W | Fasinumab 6 mg SC Q4W and Placebo IV Q8W | Fasinumab 9 mg SC Q4W and Placebo IV Q8W | Fasinumab 9 mg IV Q8W and Placebo SC Q4W
Started (Full analysis set (FAS): All randomized participants per interactive voice response system (IVRS)) | 141 | 141 | 140 | 141
Modified Intent to Treat Set (mITT) (mITT: Participants who received at least 1 dose of study drug & data up to 5 wks after last dose) | 140 | 139 | 139 | 140
Completed | 97 | 106 | 115 | 115
Not Completed | 44 | 35 | 25 | 26
Not completed — Adverse Event | 8 | 4 | 3 | 5
Not completed — Lost to Follow-up | 4 | 8 | 1 | 4
Not completed — Physician Decision | 7 | 4 | 3 | 4
Not completed — Protocol Violation | 5 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 20 | 16 | 17 | 12
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized patients per Interactive voice response system (IVRS) and was based on the treatment allocated (as randomized).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo SC Q4W and Placebo IV Q8W | Fasinumab 6 mg SC Q4W and Placebo IV Q8W | Fasinumab 9 mg SC Q4W and Placebo IV Q8W | Fasinumab 9 mg IV Q8W and Placebo SC Q4W | Total
Number analyzed (Participants) | 141 | 141 | 140 | 141 | 563
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (12.54) | 58.2 (11.29) | 56.6 (10.99) | 55.4 (10.49) | 57.1 (11.38)
Age, Customized [Number; unit: Participants]
  < 65 years | 93 | 95 | 109 | 117 | 414
  ≥ 65 years | 48 | 46 | 31 | 24 | 149
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 85 | 84 | 81 | 333
  Male | 58 | 56 | 56 | 60 | 230
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 4 | 10 | 25
  Not Hispanic or Latino | 134 | 135 | 135 | 131 | 535
  Unknown or Not Reported | 0 | 2 | 1 | 0 | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 127 | 119 | 118 | 116 | 480
  Black or African American | 13 | 19 | 19 | 21 | 72
  Asian | 1 | 2 | 2 | 1 | 6
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Other | 0 | 0 | 1 | 1 | 2
Low Back Pain Intensity Numerical Rating Scale (LBPI NRS) Baseline Score [Mean (Standard Deviation); unit: Scores on a scale] — Pre-randomization visit: Investigator recorded LBPI NRS score indicating pain intensity over past 24 hrs. per participant's report; Eligibility confirmed; LBPI NRS scores were reported by participant into electronic diary (EDiary) every day from pre-randomization to week 16; Avg. daily LBP: assessed on an 11-point numeric rating scale (NRS) defined as avg. of non-missing daily LBPI NRS scores for 7 days before, including nominal visit; Participants described avg. LBP during past 24 hrs. on a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicate higher pain. Population: Full analysis set (FAS): included all randomized patients per IVRS and was based on the treatment allocated (as randomized). Baseline number analyzed = number of participants in FAS; number analyzed here = number of participants within a specified category. EDiary NRS data were missing for some participants at Baseline.
  Scores on a scale
    number analyzed (Participants) | 140 | 139 | 140 | 141 | 560
    (all) | 6.50 (1.297) | 6.49 (1.2481) | 6.66 (1.300) | 6.45 (1.191) | 6.53 (1.267)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 16 in the Average Daily Low Back Pain Index Numeric Rating Scale (LBPI NRS) Score
Description: Average daily low back pain (LBP) was assessed on an 11-point numeric rating scale (NRS) and was defined as the average of the non-missing daily LBPI NRS scores for the 7 days before and including nominal visit. Participants described their average low back pain during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicate higher pain.
Time Frame: Baseline to Week 16
Population: Analysis performed on modified intent to treat set (mITT) included all randomized participants who received at least one dose of study drug based on the treatment allocated (as randomized) including data up to 5 weeks after the last dose of study drug. Number of participants analyzed = participants with available data for specified time point.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo SC Q4W and Placebo IV Q8W | Fasinumab 6 mg SC Q4W and Placebo IV Q8W | Fasinumab 9 mg SC Q4W and Placebo IV Q8W | Fasinumab 9 mg IV Q8W and Placebo SC Q4W
Number analyzed (Participants) | 140 | 139 | 139 | 140
Scores on a scale | -1.7 (0.23) | -2.0 (0.23) | -2.5 (0.22) | -2.4 (0.22)
Statistical Analysis 1: Comparison: Placebo SC Q4W and Placebo IV Q8W vs Fasinumab 6 mg SC Q4W and Placebo IV Q8W; Test type: Superiority; p = 0.3876, Mixed Models Analysis — Nominal p-value; Least Squares (LS) Mean Difference = -0.3, 95% CI 2-sided [-0.88 to 0.34], Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: Placebo SC Q4W and Placebo IV Q8W vs Fasinumab 9 mg SC Q4W and Placebo IV Q8W; Test type: Superiority; p = 0.0180, Mixed Models Analysis — Nominal p-value; LS Mean Difference = -0.7, 95% CI 2-sided [-1.32 to -0.12], Standard Error of Mean 0.3
Statistical Analysis 3: Comparison: Placebo SC Q4W and Placebo IV Q8W vs Fasinumab 9 mg IV Q8W and Placebo SC Q4W; Test type: Superiority; p = 0.0288, Mixed Models Analysis — Nominal p-value; LS Mean Difference = -0.7, 95% CI 2-sided [-1.26 to -0.07], Standard Error of Mean 0.3

2. Secondary Outcome: Change From Baseline to Weeks 2, 4, 8, and 12 in the Average Low Back Pain Index Numeric Rating Scale Score (LBPI NRS)
Description: as for outcome 1
Time Frame: Baseline to Weeks 2, 4, 8, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo SC Q4W and Placebo IV Q8W | Fasinumab 6 mg SC Q4W and Placebo IV Q8W | Fasinumab 9 mg SC Q4W and Placebo IV Q8W | Fasinumab 9 mg IV Q8W and Placebo SC Q4W
Number analyzed (Participants) | 140 | 139 | 139 | 140
Scores on a scale
  Change from Baseline to Week 2: number analyzed (Participants) | 136 | 133 | 135 | 138
  Change from Baseline to Week 2 | -0.9 (0.17) | -1.3 (0.17) | -1.6 (0.17) | -1.6 (0.16)
  Change from Baseline to Week 4: number analyzed (Participants) | 133 | 132 | 128 | 132
  Change from Baseline to Week 4 | -0.9 (0.17) | -1.5 (0.17) | -2.0 (0.17) | -1.9 (0.16)
  Change from Baseline to Week 8: number analyzed (Participants) | 95 | 98 | 105 | 103
  Change from Baseline to Week 8 | -1.2 (0.19) | -1.8 (0.19) | -2.3 (0.19) | -2.2 (0.19)
  Change from Baseline to Week 12: number analyzed (Participants) | 69 | 69 | 74 | 76
  Change from Baseline to Week 12 | -1.5 (0.21) | -2.0 (0.21) | -2.6 (0.21) | -2.5 (0.21)

3. Secondary Outcome: Change From Baseline to Week 16 in Roland Morris Disability Questionnaire (RMDQ) Total Score
Description: The RMDQ is a self-administered, widely used health status measure for lower back pain (LBP). It measures pain and function, using 24 items describing limitations to everyday life that can be caused by LBP. The score of the RMDQ is the total number of items checked - that is from a minimum of 0 (no disability) to a maximum of 24 (maximum disability), where lower scores indicative of better function.
Time Frame: Baseline to Week 16
Population: Analysis was performed on mITT population. Here, number of participants analyzed = participants with available data for specified time point.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo SC Q4W and Placebo IV Q8W | Fasinumab 6 mg SC Q4W and Placebo IV Q8W | Fasinumab 9 mg SC Q4W and Placebo IV Q8W | Fasinumab 9 mg IV Q8W and Placebo SC Q4W
Number analyzed (Participants) | 46 | 46 | 55 | 55
Units on a scale | -3.8 (0.54) [lower limit 0.54] | -6.0 (0.54) [lower limit 0.54] | -5.8 (0.51) [lower limit 0.51] | -6.3 (0.51) [lower limit 0.51]
Statistical Analysis 1: Comparison: Placebo SC Q4W and Placebo IV Q8W vs Fasinumab 6 mg SC Q4W and Placebo IV Q8W; Test type: Superiority; p = 0.0028, Mixed Models Analysis — Nominal p-value; LS mean difference = -2.2, 95% CI 2-sided [-3.65 to -0.77], Standard Error of Mean 0.73
Statistical Analysis 2: Comparison: Placebo SC Q4W and Placebo IV Q8W vs Fasinumab 9 mg SC Q4W and Placebo IV Q8W; Test type: Superiority; p = 0.0068, Mixed Models Analysis — Nominal p-value; LS Mean Difference = -2, 95% CI 2-sided [-3.36 to -0.54], Standard Error of Mean 0.72
Statistical Analysis 3: Comparison: Placebo SC Q4W and Placebo IV Q8W vs Fasinumab 9 mg IV Q8W and Placebo SC Q4W; Test type: Superiority; p = 0.0006, Mixed Models Analysis — Nominal p-value; LS Mean Difference = -2.5, 95% CI 2-sided [-3.88 to -1.06], Standard Error of Mean 0.72

4. Secondary Outcome: Change From Baseline to Week 16 in the Patient Global Assessment (PGA) of Low Back Pain (LBP) Score
Description: The PGA of LBP is a participant assessed 5 point Likert scale of LBP ranging from 0-5 where 1=very well; 2=well; 3=fair; 4=poor; and 5=very poor.
Time Frame: Baseline to Week 16
Population: Analysis was performed on mITT population. Here, number of participants analyzed=participants with available data for specified time point.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo SC Q4W and Placebo IV Q8W | Fasinumab 6 mg SC Q4W and Placebo IV Q8W | Fasinumab 9 mg SC Q4W and Placebo IV Q8W | Fasinumab 9 mg IV Q8W and Placebo SC Q4W
Number analyzed (Participants) | 50 | 48 | 55 | 57
Units on a scale | -0.7 (0.10) [lower limit 0.10] | -0.9 (0.10) [lower limit 0.10] | -0.8 (0.10) [lower limit 0.10] | -1.0 (0.09) [lower limit 0.09]
Statistical Analysis 1: Comparison: Placebo SC Q4W and Placebo IV Q8W vs Fasinumab 6 mg SC Q4W and Placebo IV Q8W; Test type: Superiority; p = 0.1501, Mixed Models Analysis — Nominal p-value; LS Mean Difference = -0.2, 95% CI 2-sided [-0.46 to 0.07], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo SC Q4W and Placebo IV Q8W vs Fasinumab 9 mg SC Q4W and Placebo IV Q8W; Test type: Superiority; p = 0.2603, Mixed Models Analysis — Nominal p-value; LS Mean Difference = -0.1, 95% CI 2-sided [-0.41 to 0.11], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Placebo SC Q4W and Placebo IV Q8W vs Fasinumab 9 mg IV Q8W and Placebo SC Q4W; Test type: Superiority; p = 0.0135, Mixed Models Analysis — Nominal p-value; LS Mean Difference = -0.3, 95% CI 2-sided [-0.59 to -0.07], Standard Error of Mean 0.13

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Week 36) regardless of seriousness or relationship to investigational product.
Description: Safety analysis set (SAF): All randomized participants who received any study drug (based on treatment received [as treated]). Reported AEs & deaths are treatment emergent: AEs that developed/worsened & deaths that occurred during 'treatment emergent period' (from 1st dose of study drug up to 4 wks after last dose of SC drug, or 8 wks after last dose of IV study drug, whichever is later). Reported death occurred during post-treatment follow-up period in fasinumab 6 mg SC Q4W & placebo IV Q8W arm
Groups:
- Placebo SC Q4W and Placebo IV Q8W: Participants randomized to the matching placebo subcutaneously (SC) every four weeks (Q4W) arm received SC placebo in a manner similar to the SC loading dose of the active groups (placebo loading dose) on Day 1 and then an SC injection of placebo at weeks 4, 8, and 12 for a total of 4 doses. Matching placebo intravenously (IV) every 8 weeks (Q8W) was received on Day 1 and at Week 8. Patients randomized to the 'Placebo SC Q4W and Placebo IV Q8W" treatment arm who wrongly received at least one dose of active treatment were classified in the active treatment group in the SAF.
- Fasinumab 6 mg SC Q4W and Placebo IV Q8W: Participants randomized to the fasinumab 6 mg SC Q4W arm received fasinumab 12 mg SC on Day 1 (loading dose) and then 6 mg SC (planned maintenance dose) at Weeks 4, 8, and 12 for a total of 4 doses. Matching placebo was received via intravenous (IV) infusion Q8W on Day 1 and at Week 8. Participants randomized to any of the active treatment groups receiving active fasinumab doses who wrongly received another dose of fasinumab were classified to the arm of the lowest dose of fasinumab received. For example, a participant randomized to the 'fasinumab 9 mg SC Q4W and placebo 9 mg IV Q8W' who wrongly received treatment with fasinumab 6 mg SC at least once was classified under the 'fasinumab 6 mg SC Q4W and placebo IV Q8W' treatment arm.
- Fasinumab 9 mg SC Q4W and Placebo IV Q8W: Participants randomized to the fasinumab 9 mg SC Q4W arm received 18 mg SC on day 1 (loading dose) and then 9 mg SC (planned maintenance dose) at weeks 4, 8, and 12 for a total of 4 doses. Matching placebo IV Q8W was received on Day 1 and at Week 8. Participants randomized to any of the active treatment groups receiving active fasinumab doses who wrongly received another dose of fasinumab were classified to the arm of the lowest dose of fasinumab received. For example, a participant randomized to the 'fasinumab 9 mg SC Q4W and placebo 9 mg IV Q8W' who wrongly received treatment with fasinumab 6 mg SC at least once was classified under the 'fasinumab 6 mg SC Q4W and placebo IV Q8W' treatment arm.
- Fasinumab 9 mg IV Q8W and Placebo SC Q4W: Participants randomized to the fasinumab 9 mg IV Q8W arm received IV infusions of fasinumab 9 mg on Day 1 and Week 8, for a total of 2 doses. Matching placebo SC Q4W was received on day 1 and at weeks 4, 8, and 12. Participants randomized to any of the active treatment groups receiving active fasinumab doses who wrongly received another dose of fasinumab were classified to the arm of the lowest dose of fasinumab received. For example, a participant randomized to the 'fasinumab 9 mg SC Q4W and placebo 9 mg IV Q8W' who wrongly received treatment with fasinumab 6 mg SC at least once was classified under the 'fasinumab 6 mg SC Q4W and placebo IV Q8W' treatment arm.
Arm/Group | Placebo SC Q4W and Placebo IV Q8W | Fasinumab 6 mg SC Q4W and Placebo IV Q8W | Fasinumab 9 mg SC Q4W and Placebo IV Q8W | Fasinumab 9 mg IV Q8W and Placebo SC Q4W
All-Cause Mortality (participants affected / at risk) | 0/140 | 1/139 | 0/139 | 0/140
Serious Adverse Events (participants affected / at risk) | 4/140 | 2/139 | 3/139 | 5/140
Other Adverse Events (participants affected / at risk) | 44/140 | 35/139 | 52/139 | 49/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo SC Q4W and Placebo IV Q8W (N=140) | Fasinumab 6 mg SC Q4W and Placebo IV Q8W (N=139) | Fasinumab 9 mg SC Q4W and Placebo IV Q8W (N=139) | Fasinumab 9 mg IV Q8W and Placebo SC Q4W (N=140)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo SC Q4W and Placebo IV Q8W (N=140) | Fasinumab 6 mg SC Q4W and Placebo IV Q8W (N=139) | Fasinumab 9 mg SC Q4W and Placebo IV Q8W (N=139) | Fasinumab 9 mg IV Q8W and Placebo SC Q4W (N=140)
Nausea (Gastrointestinal disorders) | 2 (4) | 4 (4) | 7 (7) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (8) | 9 (9) | 8 (9) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (22) | 15 (26) | 16 (24) | 21 (26)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0) | 4 (4) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (14) | 3 (4) | 5 (5) | 4 (7)
Headache (Nervous system disorders) | 9 (11) | 9 (9) | 9 (19) | 9 (9)
Hypoaesthesia (Nervous system disorders) | 4 (4) | 4 (4) | 7 (7) | 3 (3)
Paraesthesia (Nervous system disorders) | 4 (5) | 6 (6) | 9 (10) | 9 (9)

LIMITATIONS AND CAVEATS:
FDA placed study on partial clinical hold. Sponsor did not amend the protocol and enrollment and dosing were not resumed. However randomized participants completed all remaining study visits/procedures per protocol except for dosing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2016-08-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT02620020/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT02620020/SAP_001.pdf